CLINICAL TRIAL: NCT00513201
Title: Lyspro Insulin vs Regular Insulin in Cirrhotic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: Second University of Naples
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2007-08-08 (Estimated); Status verified 2007-08

CONDITIONS: Diabetes Mellitus; Cirrhosis
Keywords: lyspro; regular insulin; cirrhotic patients
MeSH Terms: conditions — Diabetes Mellitus; Fibrosis; Insulin Resistance | interventions — Insulin Lispro; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: lyspro
Drug: regular insulin

SUMMARY:
OBJECTIVE: To compare lispro insulin and regular insulin in the glycemic control of patients with liver cirrhosis and type 2 diabetes subjects. METHODS: 108 patients with liver cirrhosis and type 2 diabetes were randomly treated with regular insulin or lispro. After 122 weeks a cross-over was carried out and patients followed-up for 122 weeks. Then, all patients received a standard breakfast of 145 kcal following 12 U.I. of regular insulin or lispro, and C-peptide and insulin serum levels were determined over 300 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Insulin-treated diabetes mellitus and liver cirrhosis

Exclusion Criteria:

* Oral hypoglycemic agents treated diabetes mellitus
* Liver cancer

Ages: 48 Years to 67 Years | Sex: All
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Glycemic control in lyspro vs regular insulin treated patients
Glycemic control in lyspro vs regular insulin in cirrhotic patients

SECONDARY OUTCOMES:
Tolerance to treatment and reduced postprandial hypoglycemia episodes

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Torella, MD, Study Chair — University of Campania Luigi Vanvitelli
Locations (1):
- Department of Medicine, Naples, Naples, Italy